CLINICAL TRIAL: NCT05184127
Title: Open Multicenter Controlled Clinical Trial to Evaluate Safety and Efficacy of Aerosolized MIR 19 ® Inhalation in Patients With Moderate COVID-19 Who Did Not Require Treatment in the Intensive Care Unit.
Brief Title: Evaluation of Safety & Efficacy of MIR 19 ® Inhalation Solution in Patients With Moderate COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Research Center - Institute of Immunology Federal Medical-Biological Agency of Russia (Other)
Collaborators: St. Petersburg Research Institute of Vaccines and Sera (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SiCoV/KK46- 2021_CSR
Record Dates: First submitted 2022-01-07; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
Keywords: COVID-19; siRNA; SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIR 19 ® (Experimental): Study participants from experimental groups, in addition to standard COVID-19 therapy, received the MIR 19 ® (2 inhalations per day with a single dose of 1.85 or 5.55 mg at intervals of 7-8 hours for 14 days).The standard therapy in this group included symptomatic treatment without use of any etiotropic drugs such as Favipiravir, Umifenovir, Remdesivir, convalescent plasma and interferon α-2b
  Interventions: Drug: MIR 19 ®; Combination Product: Standard COVID-19 therapy
- Standard COVID-19 therapy (Active Comparator): In the comparison group, therapy was carried out in accordance with the current version of the temporary methodological recommendations of the Ministry of Health of the Russian Federation for the treatment of COVID-19 infection.The standard therapy included symptomatic treatment as well as etiotropic drugs such as Favipiravir, Umifenovir, Remdesivir, convalescent plasma and interferon α-2b. In the experimental groups treated with MIR 19 ®, the therapy included symptomatic treatment without use of any etiotropic drugs such as Favipiravir, Umifenovir, Remdesivir, convalescent plasma and interferon α-2b.
  Interventions: Combination Product: Standard COVID-19 therapy

INTERVENTIONS:
Drug: MIR 19 ® — Drug contains anti-SARS-CoV-2 siRNAs/KK-46 (peptide dendrimer) complexes for inhalation use.
  Arms: MIR 19 ®
Combination Product: Standard COVID-19 therapy — Therapy carried out in accordance with the current version of the temporary methodological recommendations of the Ministry of Health of the Russian Federation for the treatment of COVID-19 infection. This therapy included symptomatic treatment as well as etiotropic drugs such as Favipiravir, Umifenovir, Remdesivir, convalescent plasma and interferon α-2b. In the experimental groups treated with MIR 19 ®, the therapy included symptomatic treatment without use of any etiotropic drugs such as Favipiravir, Umifenovir, Remdesivir, convalescent plasma and interferon α-2b

SUMMARY:
This is Phase 2 multi-center controlled randomized study to assess the efficacy and safety of MIR 19® via 14 days of treatment of participants with symptomatic moderate COVID-19.

The purpose of this study is to evaluate the efficacy, safety and daily dose of MIR 19 ® for the treatment of the hospitalized patients with infection caused by SARS-CoV-2 (COVID-19) who did not require treatment in the intensive care unit.

Based on preclinical data studying antiviral effect of MIR 19® in vitro and in vivo (Khaitov M.R. et all 2021), the investigators hypothesized that SARS-CoV-2 inhibition with MIR 19® could potentially reduce pulmonary inflammation, thereby improving COVID-19 patient outcomes.

DETAILED DESCRIPTION:
This is Phase 2 multi-center controlled randomized study to assess the efficacy and safety of MIR 19 ® in male and female volunteers with symptomatic moderate COVID-19 who did not require treatment in the intensive care unit.

The MIR 19® is a complex of siRNA, targeting SARS-CoV-2 RNA-dependent RNA polymerase (RdRp) and peptide dendrimer KK-46.

This study involved 3 cohorts who received:

1. standard therapy which included symptomatic treatment as well as etiotropic drugs such as Favipiravir, Umifenovir, Remdesivir, convalescent plasma and interferon α-2b.
2. 3.7 mg of the MIR 19 ® via inhalation route plus standard therapy which included symptomatic treatment, without any etiotropic drugs such as Favipiravir, Umifenovir, Remdesivir, convalescent plasma and interferon α-2b.
3. 11.1 mg of the MIR 19 ® via inhalation route plus standard therapy which included symptomatic treatment, without any etiotropic drugs such as Favipiravir, Umifenovir, Remdesivir, convalescent plasma and interferon α-2b.

All subjects will undergo scheduled safety and efficacy assessments while in the clinical unit and as outpatients to the end of the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Men or non-pregnant female aged 18 to 65 years hospitalized with moderate COVID-19 infection: body temperature > 37.5 °C; respiratory rate > 22/min; shortness of breath during physical exertion; typical coronavirus-associated chest computed tomography (CT) changes (CT1- CT2); pulse oximetry levels SpO2< 95%.
2. Able to give informed consent and attend all study visits
3. Positive PCR-test for COVID-19 ≤72 hours prior to randomization
4. The patient's ability to inhale the experimental drug
5. Participants must agree to use the reliable contraception while on study medication and for posttrial contraception for 3 month

Key Exclusion Criteria:

1. Fever > 38.5°C.
2. Cough severity is less than 1 point on a 4-point scale.
3. Respiratory rate > is more than 30 / min
4. SpO2 ≤ 93%.
5. Decreased level of consciousness, agitation.
6. Unstable hemodynamics (systolic blood pressure less than 100 mmHg or diastolic blood pressure less than 60 mmHg).
7. The need to require mechanical ventilation beyond the screening/ randomization.
8. Long-term systemic corticosteroid exposure.
9. Autoimmune or inflammatory diseases (systemic / localized).
10. Positive blood tests for HIV, hepatitis B and С, syphilis.
11. Pregnancy and breast-feeding
12. Previous adverse reactions to the active substance and/or excipients included in the drug.
13. Any use of anti-viral medications or immunomodulatory agents up to 7 days before participating in the study
14. Chronic diseases of the cardiovascular system
15. Type 1 diabetes
16. The following laboratory parameters are excluded:

    Alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, total and direct bilirubin >4 x upper limit of normal (ULN);
17. Treatment with any medicine that have a pronounced effects on the blood coagulation system (expect for COVID-19 treatment), including combined oral contraceptives.
18. Treatment with any medicine that can affect cardiac conduction
19. Participation in other investigational drug or device clinical trials within 90 days prior to screening.
20. History of alcohol, drug or chemical abuse.
21. Mental illness.
22. Receipt of plasma from a person who recovered from COVID-19 (convalescent plasma) up to 14 days before participating in the study, vaccination against SARS-CoV-2 , the need for extracorporeal membrane oxygenation.
23. Any conditions that, according to the researcher's, may be a contraindication to the participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Relief of fever | Within 14 days
  Reduction in axillary temperature below 37 °C without antipyretic drugs use
Respiratory rate | Within 14 days
  Respiratory rate ≤ 22 per minute
Oxygen saturation | Within 14 days
  SpO2 > 94%
Severity of cough | Within 14 days
  Severity in a patient's cough no more than 1 point on a four-point scale

CONTACTS AND LOCATIONS:
Locations (1):
- NRC Institute of Immunology FMBA, Moscow, Russia

REFERENCES:
- [Derived] Khaitov M, Nikonova A, Kofiadi I, Shilovskiy I, Smirnov V, Elisytina O, Maerle A, Shatilov A, Shatilova A, Andreev S, Sergeev I, Trofimov D, Latysheva T, Ilyna N, Martynov A, Rabdano S, Ruzanova E, Savelev N, Pletiukhina I, Safi A, Ratnikov V, Gorelov V, Kaschenko V, Kucherenko N, Umarova I, Moskaleva S, Fabrichnikov S, Zuev O, Pavlov N, Kruchko D, Berzin I, Goryachev D, Merkulov V, Shipulin G, Udin S, Trukhin V, Valenta R, Skvortsova V. Treatment of COVID-19 patients with a SARS-CoV-2-specific siRNA-peptide dendrimer formulation. Allergy. 2023 Jun;78(6):1639-1653. doi: 10.1111/all.15663. Epub 2023 Feb 14. PMID 36721963